CLINICAL TRIAL: NCT04989231
Title: An Open and Observational Phase Ⅳ Clinical Trial to Evaluate the Immunity Persistence of Sabin Inactivated Poliovirus Vaccine (Vero Cell) After Four Doses
Brief Title: An Immunity Persistence Study of Sabin Inactivated Poliovirus Vaccine(Vero Cell) After Four Doses
Status: Completed | Type: Observational
Sponsor: Sinovac Biotech Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: PRO-sIPV-3003
Record Dates: First submitted 2021-07-14; First posted 2021-08-04 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2021-10

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The serum samples of this study will be only used for neutralizing antibody detection to evaluate immune persistence, and the use of other studies requires the consent of the subject's guardian and the approval of the ethics committee. Except for the serum submitted for testing, the remaining serum will be stored at the study site until the end of the study, and will be handed over to the sponsor for destruction according to the established SOP.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Experimental Group: Subjects who have received 4 doses of the experimental vaccine (including subjects at the age of 4 years (48 to 54 months) and 5 years (78 to 84 months) after the last vaccination ) will be collected venous blood about 3.0ml.
  Interventions: Biological: Investigational sIPV
- Control Group: Subjects who have received 4 doses of control vaccine (including subjects at the age of 4 years (48 to 54 months) and 5 years (78 to 84 months) after the last vaccination ) will be collected venous blood about 3.0ml.
  Interventions: Biological: Control IPV

INTERVENTIONS:
Biological: Investigational sIPV — Three intramuscular injections of the investigational vaccine (0.5 ml) at 0 month ,1 month and 2 months respectively; Single intramuscular injection of the investigational vaccine (0.5 ml) at 18 months
  Groups: Experimental Group
Biological: Control IPV — Three intramuscular injections of the control vaccine (0.5 ml) at 0 month ,1 month and 2 months respectively;Single intramuscular injection of the control vaccine (0.5ml) at 18 months
  Groups: Control Group

SUMMARY:
This is an open and observational follow-up clinical trial based on the previous Phase III clinical trial of Sabin Inactivated Poliovirus Vaccine manufactured by Sinovac Biotech Co. , the purpose of this study is to evaluate the immunity persistence of sIPV in infants after 4 doses of vaccination.

DETAILED DESCRIPTION:
This study is an open and observational follow-up clinical trial based on the previous Phase III clinical trial of Sabin Inactivated Poliovirus Vaccine.The purpose of this study is to evaluate the immunity persistence of sIPV in infants after 4 doses of vaccination.A total of at least 450 subjects who have received 4 doses of the experimental vaccine or control vaccine will be enrolled,about 3.0ml of venous blood will be collected from each enrolled subject at the age of 4 years (48 to 54 months) and 5 years (78 to 84 months) after the last vaccination, respectively,and the serum will be separated for neutralizing antibody detection.The antibody levels of the experimental vaccine group and the control vaccine group will be compared to evaluate the immunity persistence of sIPV.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have received 4 doses of experimental vaccine or control vaccine in phase Ⅲ clinical trials

Exclusion Criteria:

* History of vaccination of other vaccine with poliovirus antigenic components except that of phaseⅢ clinical trial.

Ages: 48 Months to 84 Months | Sex: All
Age Groups: Child
Study Population: A total of at least 450 subjects will be enrolled, subjects should meet the inclusion criteria :Subjects who have received 4 doses of experimental vaccine or control vaccine in phase Ⅲ clinical trials and subjects should not meet the exclusion criteria:history of vaccination of other vaccine with poliovirus antigenic components except that of phaseⅢ clinical trial.
Sampling Method: Probability Sample
Enrollment: 450 (Actual)
Dates: Start 2021-09-09 (Actual); Primary Completion 2022-12-25 (Actual); Study Completion 2022-12-25 (Actual)

PRIMARY OUTCOMES:
All of participants with seroconversion rates of the neutralizing antibody of each group at the observation point wich at the age of 4 years (48 to 54 months) will be assessed | At the age of 4 years (48 to 54 months) after the vaccination of the experimental vaccine or control vaccine
  About 3.0ml of venous blood will be collected from all of the subjects at the age of 4 years (48 to 54 months) and all of the participants with seroconversion rates of the neutralizing antibody at the observation point wich at the age of 4 years (48 to 54 months) will be compared to evaluate the immunity persistence of SIPV.
All of participants with seroconversion rates of the neutralizing antibody of each group at the observation point wich in 5 years (78 to 84 months) after the last vaccination will be assessed | In 5 years (78 to 84 months) after the last vaccination of the experimental vaccine or control vaccine
  About 3.0ml of venous blood will be collected from all of the subjects in 5 years (78 to 84 months) after the last vaccination and all of the participants with seroconversion rates of the neutralizing antibody at the observation point which in 5 years (78 to 84 months) after the last vaccination will be compared to evaluate the immunity persistence of SIPV.

SECONDARY OUTCOMES:
All of participants with geometric mean titer (GMT) of each group at the observation point wich at the age of 4 years (48 to 54 months) will be assessed | At the age of 4 years (48 to 54 months)
  All of participants with geometric mean titer (GMT) in experimental group and control group at the observation point wich at the age of 4 years (48 to 54 months) will be compared to evaluate the immunity persistence of SIPV.
All of participants with geometric mean titer (GMT) of each group at the observation point wich in 5 years (78 to 84 months) after the last vaccination will be assessed | In 5 years (78 to 84 months) after the last vaccination of the experimental vaccine or control vaccine
  All of participants with geometric mean titer (GMT) in experimental group and control group at the observation point wich in 5 years (78 to 84 months) after the last vaccination of the experimental vaccine or control vaccine will be compared to evaluate the immunity persistence of SIPV.

CONTACTS AND LOCATIONS:
Overall Officials: Hongxing Pan, Master, Principal Investigator — Jiangsu Provincial Center for Disease Prevention and Control
Locations (1):
- Pizhou county Center for Disease Control and Prevention, Pizhou, Jiangsu, China

REFERENCES:
- [Derived] Chu K, Li Y, Yu D, Song Y, Liu S, Xue F, Shan Y, Meng W, Pan H. Immunogenicity and immune persistence in 4-year-old children completing four doses of Sabin strain or wild strain inactivated poliovirus vaccine: A phase IV, open-labeled, parallel-controlled observational study. Vaccine. 2023 May 22;41(22):3467-3471. doi: 10.1016/j.vaccine.2023.03.012. Epub 2023 Apr 29. PMID 37127526